CLINICAL TRIAL: NCT04021927
Title: Development of a Neonatal Jaundice Treatment Accelerator by Redirection of Unused Light During Phototherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn by funding organization with no participants enrolled
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR194709
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Jaundice; Jaundice, Neonatal
MeSH Terms: conditions — Jaundice; Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ring Phototherapy (Experimental): The product will be an open-faced ring device with an angular reflective surface that redirects unused light sideways onto the neonate's body illuminating previously unexposed regions where treatable bilirubin exists while protecting the baby from head roll with an inner transparent corral. This device is superior to current PT devices because it converts existing waste light into treatment efficacy while integrating into existing single overhead lamp systems avoiding the purchase of secondary devices that are expensive and create hospital system complexity and inefficiency issues.
  Interventions: Device: Ring Phototherapy

INTERVENTIONS:
Device: Ring Phototherapy — The product will be an open-faced ring device with an angular reflective surface that redirects unused light sideways onto the neonate's body illuminating previously unexposed regions where treatable bilirubin exists while protecting the baby from head roll with an inner transparent corral. This device is superior to current PT devices because it converts existing waste light into treatment efficacy while integrating into existing single overhead lamp systems avoiding the purchase of secondary devices that are expensive and create hospital system complexity and inefficiency issues.

SUMMARY:
This is a descriptive prospective study of safety and efficacy of the reflective PT ring device. Neonates with an elevated total serum bilirubin (TSB) meeting PT criteria per their clinician during hospital admission will be eligible for enrollment after informed parental consent.

DETAILED DESCRIPTION:
Neonatal jaundice (NNJ) continues to be a significant global problem affecting over 80% of neonates while severe neonatal jaundice affects at least 481,000 neonates annually. Jaundice and jaundice related complications like Kernicterus Spectrum Disorder (KDS) are gaining recognition among the world's health policy leaders as an important area for further research and development. The long-term sequelae of KSD include choreoathetoid cerebral palsy, sensorineural hearing loss, and upward gaze palsy. KSD is irreversible resulting in a lifetime of physical, emotional, social and economic challenges. Access to cost-effective methods of improving pediatric jaundice care along with improved circumferential (full body) illumination technologies is an affirmed objective of the AAP (American Academy of Pediatrics). The investigators hypothesize that unused therapy light (irradiance) surrounding the neonate using an existing single-lamp bank phototherapy (PT) device is sufficient in quantity and if redirected onto the patients untreated or poorly illuminated skin surfaces, it will accelerate metabolism and excretion of bilirubin. This PT ring device redirects unused phototherapy light sideways onto the neonate body using an open-faced ring approach. The technology will illuminate previously unexposed and poorly exposed skin regions where treatable bilirubin exists. The device is superior to current PT devices in that it converts existing waste light into treatment efficacy while integrating into existing overhead lamp systems offsetting the purchase of secondary devices that are often unaffordable and create hospital complexity, cost and inefficiency issues. A further benefit of the device will be reduced ambient blue-light spillover in patient care areas, an ongoing concern for medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Males or female neonates greater than or equal to 35 weeks gestational age
* Elevated total serum bilirubin levels meeting PT criteria in the first 7 days of life

Exclusion Criteria:

* Neonates, who are mechanically ventilated
* Neonates requiring continuous positive airway pressure
* Neonates with a history of apnea, bradycardia
* Patients with known cyanotic heart disease
* Patients experiencing temperature instability or desaturation episodes in 24hr prior to enrollment will be excluded.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Safety of Reflective Ring PT Device: umber of participants who experience fluctuations of body temperature | Entirety of hospital admission, approximately 5 days
  Number of participants who experience fluctuations of body temperature outside the normal range during treatment
Safety of Reflective Ring PT Device: Number of participants who experience apnea | Entirety of hospital admission, approximately 5 days
  Number of participants who experience apnea during treatment
Safety of Reflective Ring PT Device: Number of participants who experience a bradycardic episode | Entirety of hospital admission, approximately 5 days
  Number of participants who experience a bradycardic episode during treatment
Safety of Reflective Ring PT Device: Number of participants who experience an episode of oxygen desaturation | Entirety of hospital admission, approximately 5 days
  Number of participants who experience an episode of oxygen desaturation during treatment

SECONDARY OUTCOMES:
Efficacy: Percent of Participants with Normal Serum Bilirubin Concentrations | Entirety of hospital admission, approximately 5 days
  Percentage of participants who achieve normal serum bilirubin concentrations during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No